CLINICAL TRIAL: NCT06188624
Title: A Phase I Clinical Study of TQB2922 for Injection in Patients With Advanced Cancers
Brief Title: Clinical Trial of TQB2922 for Injection in Patients With Advanced Cancers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2922-I-01
Record Dates: First submitted 2023-12-19; First posted 2024-01-03 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-03

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2922 for injection (Experimental): TQB2922 for injection, 28 days as a treatment cycle
  Interventions: Drug: TQB2922 for injection

INTERVENTIONS:
Drug: TQB2922 for injection — TQB2922 for injection is administrated to patients with advanced cancers, 28 days as a treatment cycle

SUMMARY:
This is a Phase I study to evaluate the safety, tolerability, and efficacy of TQB2922 for injection in subjects with advanced cancers

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily join this study, sign the informed consent form, and have good compliance；
* Age: 18-75 years; Eastern Cooperative Oncology Group (ECOG) score: 0-1 ; Expected survival of more than 3 months；
* Histologically or cytologically diagnosed with advanced cancers;
* Subjects with advanced malignancies who have failed standard therapy or lack effective treatment;
* Major organs are functioning well;
* Female and male subjects of childbearing potential should agree to practice contraception during the study and until 6 months after the completion of the study.

Exclusion Criteria:

* Current concomitant or ever presented with other malignancies within 2 years prior to the first dose;
* Unresolved toxicity of Grade 1 or above according to CTCAE due to any prior anti-tumor therapy;
* Significant surgical treatment, biopsy, or significant traumatic injury within 28 days prior to the first dose;
* Long-term unhealed wounds or fractures
* Cerebrovascular accident (including transient ischemic attack, intracerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism within 6 months prior to the first dose;
* A history of psychotropic drug abuse and cannot be abstained, or have a mental disorder;
* Subjects with any severe and/or uncontrolled disease;
* History of live attenuated vaccination within 2 weeks prior to the first dose or planned live attenuated vaccination during the study;
* Previous history of unexplained severe allergies, hypersensitivity to monoclonal antibodies or exogenous human immunoglobulins, or hypersensitivity to TQB2922 for injection or its excipients;
* According to the judgment of the investigator, there are concomitant diseases that seriously endanger the safety of the patients or affect the completion of the study, or subjects who are considered to be unsuitable for enrollment for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | During the first treatment cycle (28 days).
  DLT is defined as toxicities that meet pre-defined severity criteria according to the NCI CTCAE (National Cancer Institute Common Terminology Criteria for Adverse Events) v5.0 toxicity assessment criteria, and assessed as having a suspected relationship to study drug that occurred.
Maximum tolerated dose (MTD) | During the first treatment cycle (28 days).
  MTD is defined as the highest dose at which dose-limiting toxicity (DLT) occurred in less than 33% of patients.
Adverse events (AEs) rate | From date of the first dose until 30 days after last dose or start with new anti-tumor treatment, whichever comes first.
  The occurrence rate of all AEs during treatment
Adverse events (AEs) severity | From date of the first dose until 30 days after last dose or start with new anti-tumor treatment, whichever comes first.
  The severity of all AEs occured during treatment

SECONDARY OUTCOMES:
Half-life (T1/2) | Pre-dose and 5 minutes post-dose on Cycle 1 Day 1, 8, 15, 22 and Cycle 2 Day 1; Pre-dose on Day 15 Cycle 2; 2, 6, 24, 72 hours after dose on Cycle 1 Day 1; 6, 24, 72, 128 hours after dose on Cycle 2 Day 1. Each cycle is 28 days.
  Terminal half-life (T1/2) after administration
The area under the curve (AUC) | Pre-dose and 5 minutes post-dose on Cycle 1 Day 1, 8, 15, 22 and Cycle 2 Day 1; Pre-dose on Day 15 Cycle 2; 2, 6, 24, 72 hours after dose on Cycle 1 Day 1; 6, 24, 72, 128 hours after dose on Cycle 2 Day 1. Each cycle is 28 days.
  The area under the curve (AUC) of blood concentration-time of TQB2922.
Apparent plasma clearance (CL) | Pre-dose and 5 minutes post-dose on Cycle 1 Day 1, 8, 15, 22 and Cycle 2 Day 1; Pre-dose on Day 15 Cycle 2; 2, 6, 24, 72 hours after dose on Cycle 1 Day 1; 6, 24, 72, 128 hours after dose on Cycle 2 Day 1. Each cycle is 28 days.
  Apparent plasma clearance of TQB2922.
Apparent volume of distribution (Vz) | Pre-dose and 5 minutes post-dose on Cycle 1 Day 1, 8, 15, 22 and Cycle 2 Day 1; Pre-dose on Day 15 Cycle 2; 2, 6, 24, 72 hours after dose on Cycle 1 Day 1; 6, 24, 72, 128 hours after dose on Cycle 2 Day 1. Each cycle is 28 days.
  The ratio of the amount of TQB2922 in the body to the blood concentration
Minimum concentration (Cmin) | Pre-dose and 5 minutes post-dose on Cycle 1 Day 1, 8, 15, 22 and Cycle 2 Day 1; Pre-dose on Day 15 Cycle 2; 2, 6, 24, 72 hours after dose on Cycle 1 Day 1; 6, 24, 72, 128 hours after dose on Cycle 2 Day 1. Each cycle is 28 days.
  Minimum observed concentration (Cmin) of TQB2922
Objective response rate (ORR) | Up to 2 years.
  The percentage of patients with complete response (CR) or partial response (PR) assessed by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1.
Duration of response (DOR) | Up to 2 years.
  The time from first documented response to documented disease progression.
Progression-free survival (PFS) | Up to 2 years.
  The time from the first dose of TQB2922 to the first occurrence of disease progression or death from any cause.
Immunogenicity of TQB2922 | From the time of informed consent to 90 days after the last dose.
  Immunogenicity of TQB2922 is assessed according to the incidence of anti-drug antibody (ADA).

CONTACTS AND LOCATIONS:
Locations (17):
- China (17):
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The first affiliated hospital of Guangzhou medical university, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Henan Provincine People's Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Affiliated Zhongshan Hospital of Dalian University, Dalian, Liaoming
  - Department of Medical Oncology, The First Hospital of China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Affiliated Hospital of North Sichuan Medical College, Nanchong, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Yunnan Cancer Hospital, Kunming, Yunnan